CLINICAL TRIAL: NCT06346990
Title: The Effect of Listening to Holy Quran Recital on the Incidence of Delirium Post-CABG: A Randomized Control Trial
Brief Title: The Effect of Listening to Holy Quran Recital on the Incidence of Delirium Post-CABG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mohannad Aburuz, Professor of Critical Care Nursing, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Faculty 2023-2024-2-2
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft Surgery; Delirium, Postoperative
Keywords: Delirium; length of stay
MeSH Terms: conditions — Coronary Artery Disease; Emergence Delirium; Delirium

STUDY DESIGN:
Intervention Model Description: There are two groups in this study. The intervention group and the control group. For the control group, patients are receiving routine care . For the intervention group, after patients were (1) extubated, (2) hemodynamically stable, and (3) negatively rated on primary CAM-ICU, they receive holy Quran recital for four days. Typically, the second, third, fourth- and fifth-days following CABG. The daily sessions were done at 2 PM and 8 PM for 20 minutes each. We choose these times based on the nurses' recommendations about the minimal interruptions from physician rounds and family visits. The selection of Surah Al-Rahman was based on the widespread belief that it is among the most melodic and calming passages in the Quran, especially when recited by the well-known reciter Qari AbdulBasit. 1,5,40 The listening was done using one-use headphones on an iPad. The intervention was discontinued if the participant developed delirium
Who Masked: Outcomes Assessor
Masking Description: Taking into consideration that this was a RCT, blinding the participants was not possible. However, data collectors and data analyzer were blinded. Directly after the intervention, each day at 3pm and 9 pm, the participants were evaluated for development of delirium by the Research assistant how do not know in which group was the participant allocated, and if the result was positive the intervention was discontinued.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group/ Holy Quran Recital (Experimental): For the intervention group, after patients were (1) extubated, (2) hemodynamically stable, and (3) negatively rated on primary CAM-ICU, they received holy Quran recital for four days. Typically, the second, third, fourth- and fifth-days following CABG. The daily sessions were done at 2 PM and 8 PM for 20 minutes each. We choose these times based on the nurses' recommendations about the minimal interruptions from physician rounds and family visits. The selection of Surah Al-Rahman was based on the widespread belief that it is among the most melodic and calming passages in the Quran, especially when recited by the well-known reciter Qari AbdulBasit. 1,5,40 The listening was done using one-use headphones on an iPad. The intervention was discontinued if the participant developed delirium.
  Interventions: Other: Holy Quran Recital
- The control group (No Intervention): For the control group, routine post-operative care was done

INTERVENTIONS:
Other: Holy Quran Recital — Holy Quran recital for four days. Typically, the second, third, fourth- and fifth-days following CABG. The daily sessions were done at 2 PM and 8 PM for 20 minutes each
  Arms: The intervention group/ Holy Quran Recital

SUMMARY:
This study is planned to check the effect of holy Quran recital on the development of delirium after conronary artery bypass graft surgery (CABG). Different studies have been done before about the effects of non-pharmacological intervention on delirium after CABG, howvere, none was designed specifically to check the effect of Holy Qoyran on this outcome.

DETAILED DESCRIPTION:
Coronary artery disease is a very common cardiovascular disease nationwide. Coronary artery bypass graft surgery (CABG) is a surgical treatment for coronary artery disease. This surgery has positive outcomes for the patients compared to other revascularization procedures including lower levels of re-infarctions, better quality of life, extend patients' lives and reduction of revascularization procedures. Despite these benefits, CABG is a major surgery that has its own risks and complications, like bleeding, wound infection, extended use of mechanical ventilation, cardiac dysthymias, stroke, pulmonary edema, death, and development of post-operative delirium. The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) describes delirium as a transient mental syndrome that is characterized by three main symptoms: "(a) Disturbance in attention (i.e., reduced ability to direct, focus, sustain, and shift attention) and awareness (reduced orientation to the environment), (b) The disturbance develops over a short period of time (usually hours to a few days), represents an acute change from baseline attention and awareness, and tends to fluctuate in severity during the course of a day, (c) An additional disturbance in cognition (e.g. memory deficit, disorientation, language, visuospatial ability, or perception)." There is also a need for evidence from physical exam and laboratory findings that these changes are not due to other conditions like drug abuse, withdrawal symptoms, or the use of medications.9 Delirium is a common complication after CABG with high incidence rates ranging from 3% to 75%. These high rates are linked to a number of negative outcomes, including self-extubation, respiratory failure, sternal instability, an extended hospital stay, higher (readmissions, medical expenses, and mortality rates) and lower quality of life. Even though delirium is common and has detrimental clinical effects, medical professionals and staff frequently fail to recognize it. According to earlier research, between 32% and 84% of delirium cases go undetected by medical professionals. Most of delirium cases occur after major and long surgeries like CABG, not after minor surgeries. These results indicate that the pathophysiology of postoperative delirium may be significantly influenced by anxiety, stress and depressive responses brought on by surgical stimulation has been reported that stress, anxiety and depression were high in the per-operative period and were associated negative outcomes as increased length of stay and occurrence delirium. Primary prevention of delirium entails reducing effective risk factors such environmental interventions, while secondary prevention involves early diagnosis. Increasing or lowering environmental stimulation, medicine, and music therapy are some strategies to lower the frequency of delirium. Fortunately, delirium is a sickness that can be avoided. Instead of treating this illness, researchers have recently concentrated more on risk factor identification and prevention. Therefore, investigations involving medications like melatonin, reduction of sedative medications as benzodiazepines, and surgical methods were conducted with the aim of preventing these postoperative morbidities; however, the results have been inconclusive.

Consequently, non-pharmacological intervention to control delirium after CABG were studied like the use of music and education. These non-pharmacological interventions work through the hypothesis that they will regulate the effect of anxiety, stress and depression resulting in reducing heart rate, blood pressure, and pro-inflammatory cytokines. In addition, previous studies showed a connection between non-pharmacological interventions and reduction of postoperative pain, and serum cortisol levels which in turn reduced the occurrence of delirium. However, none of these studies was designed specifically to check the effect of listing to Holy Quran on the incidence of delirium post CABG, which might be working through the same mechanism. Among patients how did CABG, previous studies demonstrated that holy Quran audio therapy was significantly associated with reduction of anxiety and depressive symptoms.1,36 Moreover, listening to holy Quran recital significantly decreased pain and length of stay. Also, with regard to patients with heart problems other than CABG, Quran audio therapy has been shown to reduce anxiety before cardiac catheterization procedures, and enhance sleep quality following other cardiac surgeries. Research questions: (1) what is the incidence of delirium post CABG, (2) what is the effect of listing to holy Quran on the incidence of delirium post CABG, (3) what is the effect of listing to holy Quran on the length of stay post CABG, and (4) what is the effect of delirium on the length of stay (LoS) post CABG.

ELIGIBILITY:
Inclusion Criteria:.

* 18 years old and older;
* undergone elective CABG surgery;
* hemodynamically stable during interventions and interviews;
* signed an informed consent
* Exclusion Criteria:
* Developed delirium before the intervention based on Confusion Assessment Method for the Intensive Care Unit (CAM-ICU);
* Had a history of liver cirrhosis, kidney failure, stroke, dementia, or psychiatric problems;
* On anti-antipsychotic medications; or
* Received treated with ketamine or midazolam in the operating room or benzodiazepines, haloperidol, and propofol in the intensive care unit (ICU), as they are known to increase susceptibility for hallucination and delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Delirium | Within one week after the operation
  The effect of holy quran recital on the incidence of delirium

SECONDARY OUTCOMES:
Length of stay-ICU | Within one week after the operation
  The effect of holy quran recital on the length of stay in the ICU
Length of stay-hospital | Within two week after the operation
  The effect of holy quran recital on the length of stay in the hospital

IPD SHARING:
Plan to Share IPD: Undecided